CLINICAL TRIAL: NCT05575791
Title: Evaluation of Preoperative Acceptance of Proactive Palliative Care Intervention
Acronym: iCare
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Treskatsch, Univ.-Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA1/292/20
Record Dates: First submitted 2022-02-21; First posted 2022-10-12 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Cancer; Heart Failure; Chronic Obstructive Pulmonary Disease; Postoperative Complications
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Advances in medicine have led to an increased life expectancy even with complex disease courses of malignant diseases.

This leads to frequent critical situations for patients and high risk surgical interventions. The majority of patients and their practitioners are not prepared for the consequences of a complex and possibly fatal course.

Palliative medicine makes it possible to anticipate the further course of the disease. As a result, palliative medicine has become increasingly important. The beginning of palliative medical interventions has extended from accompaniment limited to the dying phase to earlier phases of the disease.

An early integration of palliative medicine showed a positive effect on the quality of life, the degree of depression and survival in patients suffering from cancer, for example. Furthermore, patients were more able to accept a change in therapy goal at the end of life. Similar results were shown for patients with a non-malignant severe disease such as COPD or heart failure.

What needs further investigating is how to adequately screen and identify the patient populations who could benefit from early palliative care, so that they are prepared for potentially critical and life-threatening situations.

The investigator's objective is therefore whether the Anesthesiology Outpatient Clinic is a suitable screening location for initiating early integrated palliative care for patients with a serious, life-shortening illness and a high perioperative risk.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* one elective operation with medium or high cardiac risk

And in addition at least one of the following criteria:

* serious comorbidity pulmonary: Emphysema and / or COPD >= 2 after GOLD cardiac: NYHA > = 2
* and / or a metastatic malignancy
* ASA physical status classification >= 3 and pre-frail or frail

Exclusion Criteria:

* legal care
* Emergency operation
* any reasons which contradict inclusion in studies , e.g. cognitive deficit and lack of language skills
* Pregnant / breastfeeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected out of the population consulted at the anesthesiology outpatient clinic of the University hospital Berlin - Charite.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Acceptance of the preoperative palliative counseling offer | through study completion, an average of 1 year
  Percentage of patients who accept the palliative counseling offer in relation to the total number of patients identified in the screening of the anesthesia outpatient clinic

SECONDARY OUTCOMES:
Advance planning documents | through study completion, an average of 1 year
  Percentage of patients who, as a result of the palliative medical consultation offer, create or want to create a living will or power of attorney
Postoperative palliative counseling | through study completion, an average of 1 year
  Percentage of patients who would like further palliative medical advice postoperatively
Acceptance of the preoperative palliative counseling offer depending on the underlying disease | through study completion, an average of 1 year
  Percentage of patients with and without a malignant disease who accept the counseling offer
Therapy target decision-making situations | through study completion, an average of 1 year
  Percentage of patients in whom a decision to limit therapy occurs in the postoperative course
Gender difference | through study completion, an average of 1 year
  Percentage of female patients who accept the counseling offer in relation to male patients
Therapy goal decisions postoperatively | through study completion, an average of 1 year
  Percentage of patients who do not accept the offer of counseling and who have difficult therapy goal decisions postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and operative intensive Care, Campus Benjamin Franklin, Charité - University Hospital Berlin, Steglitz, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Vanbutsele G, Pardon K, Van Belle S, Surmont V, De Laat M, Colman R, Eecloo K, Cocquyt V, Geboes K, Deliens L. Effect of early and systematic integration of palliative care in patients with advanced cancer: a randomised controlled trial. Lancet Oncol. 2018 Mar;19(3):394-404. doi: 10.1016/S1470-2045(18)30060-3. Epub 2018 Feb 3. PMID 29402701
- [Background] Vanbutsele G, Van Belle S, Surmont V, De Laat M, Colman R, Eecloo K, Naert E, De Man M, Geboes K, Deliens L, Pardon K. The effect of early and systematic integration of palliative care in oncology on quality of life and health care use near the end of life: A randomised controlled trial. Eur J Cancer. 2020 Jan;124:186-193. doi: 10.1016/j.ejca.2019.11.009. Epub 2019 Dec 5. PMID 31812934
- [Background] Maltoni M, Scarpi E, Dall'Agata M, Zagonel V, Berte R, Ferrari D, Broglia CM, Bortolussi R, Trentin L, Valgiusti M, Pini S, Farolfi A, Casadei Gardini A, Nanni O, Amadori D; Early Palliative Care Italian Study Group (EPCISG). Systematic versus on-demand early palliative care: results from a multicentre, randomised clinical trial. Eur J Cancer. 2016 Sep;65:61-8. doi: 10.1016/j.ejca.2016.06.007. Epub 2016 Jul 26. PMID 27472648
- [Background] Haun MW, Estel S, Rucker G, Friederich HC, Villalobos M, Thomas M, Hartmann M. Early palliative care for adults with advanced cancer. Cochrane Database Syst Rev. 2017 Jun 12;6(6):CD011129. doi: 10.1002/14651858.CD011129.pub2. PMID 28603881
- [Background] Higginson IJ, Bausewein C, Reilly CC, Gao W, Gysels M, Dzingina M, McCrone P, Booth S, Jolley CJ, Moxham J. An integrated palliative and respiratory care service for patients with advanced disease and refractory breathlessness: a randomised controlled trial. Lancet Respir Med. 2014 Dec;2(12):979-87. doi: 10.1016/S2213-2600(14)70226-7. Epub 2014 Oct 29. PMID 25465642
- [Background] Hauptman PJ, Havranek EP. Integrating palliative care into heart failure care. Arch Intern Med. 2005 Feb 28;165(4):374-8. doi: 10.1001/archinte.165.4.374. PMID 15738365
- [Background] Zhou K, Mao Y. Palliative care in heart failure : A meta-analysis of randomized controlled trials. Herz. 2019 Aug;44(5):440-444. doi: 10.1007/s00059-017-4677-8. Epub 2018 Feb 21. PMID 29468259
- [Background] Siouta N, Heylen A, Aertgeerts B, Clement P, Van Cleemput J, Janssens W, Menten J. Early integrated palliative care in chronic heart failure and chronic obstructive pulmonary disease: protocol of a feasibility before-after intervention study. Pilot Feasibility Stud. 2019 Feb 21;5:31. doi: 10.1186/s40814-019-0420-y. eCollection 2019. PMID 30834140
- [Background] Brumley R, Enguidanos S, Jamison P, Seitz R, Morgenstern N, Saito S, McIlwane J, Hillary K, Gonzalez J. Increased satisfaction with care and lower costs: results of a randomized trial of in-home palliative care. J Am Geriatr Soc. 2007 Jul;55(7):993-1000. doi: 10.1111/j.1532-5415.2007.01234.x. PMID 17608870
- [Background] Ma J, Chi S, Buettner B, Pollard K, Muir M, Kolekar C, Al-Hammadi N, Chen L, Kollef M, Dans M. Early Palliative Care Consultation in the Medical ICU: A Cluster Randomized Crossover Trial. Crit Care Med. 2019 Dec;47(12):1707-1715. doi: 10.1097/CCM.0000000000004016. PMID 31609772
- [Background] Yefimova M, Aslakson RA, Yang L, Garcia A, Boothroyd D, Gale RC, Giannitrapani K, Morris AM, Johanning JM, Shreve S, Wachterman MW, Lorenz KA. Palliative Care and End-of-Life Outcomes Following High-risk Surgery. JAMA Surg. 2020 Feb 1;155(2):138-146. doi: 10.1001/jamasurg.2019.5083. PMID 31895424
- [Background] Cancer Control: Knowledge into Action: WHO Guide for Effective Programmes: Module 5: Palliative Care. Geneva: World Health Organization; 2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK195248/ PMID 24716263
- [Background] Chan R, Ueno R, Afroz A, Billah B, Tiruvoipati R, Subramaniam A. Association between frailty and clinical outcomes in surgical patients admitted to intensive care units: a systematic review and meta-analysis. Br J Anaesth. 2022 Feb;128(2):258-271. doi: 10.1016/j.bja.2021.11.018. Epub 2021 Dec 17. PMID 34924178
- [Background] Morgeli R, Wollersheim T, Spies C, Balzer F, Koch S, Treskatsch S. [How to Reduce the Rate of Postoperative Complications in Frail Patients?]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2017 Nov;52(11-12):785-797. doi: 10.1055/s-0043-104685. Epub 2017 Nov 20. German. PMID 29156482
- [Background] Birkelbach O, Morgeli R, Balzer F, Olbert M, Treskatsch S, Kiefmann R, Muller-Werdan U, Reisshauer A, Schwedtke C, Neuner B, Spies C. [Why and How Should I Assess Frailty? A Guide for the Preoperative Anesthesia Clinic]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2017 Nov;52(11-12):765-776. doi: 10.1055/s-0043-104682. Epub 2017 Nov 20. German. PMID 29156481
- [Background] Birkelbach O, Morgeli R, Spies C, Olbert M, Weiss B, Brauner M, Neuner B, Francis RCE, Treskatsch S, Balzer F. Routine frailty assessment predicts postoperative complications in elderly patients across surgical disciplines - a retrospective observational study. BMC Anesthesiol. 2019 Nov 7;19(1):204. doi: 10.1186/s12871-019-0880-x. PMID 31699033
- [Background] de Heer G, Saugel B, Sensen B, Rubsteck C, Pinnschmidt HO, Kluge S. Advance Directives and Powers of Attorney in Intensive Care Patients. Dtsch Arztebl Int. 2017 Jun 5;114(21):363-370. doi: 10.3238/arztebl.2017.0363. PMID 28625275
- [Background] Leder N, Schwarzkopf D, Reinhart K, Witte OW, Pfeifer R, Hartog CS. The Validity of Advance Directives in Acute Situations. Dtsch Arztebl Int. 2015 Oct 23;112(43):723-9. doi: 10.3238/arztebl.2015.0723. PMID 26568176
- [Background] Schoffner M, Schmidt KW, Benzenhofer U, Sahm S. [Living wills under close scrutiny: Medical consultation is indispensable]. Dtsch Med Wochenschr. 2012 Mar;137(10):487-90. doi: 10.1055/s-0031-1298998. Epub 2012 Feb 28. German. PMID 22374658
- [Background] Pfirstinger J, Kattner D, Edinger M, Andreesen R, Vogelhuber M. The impact of a tumor diagnosis on patients' attitudes toward advance directives. Oncology. 2014;87(4):246-56. doi: 10.1159/000363508. Epub 2014 Aug 15. PMID 25139124
- [Background] Urman RD, Gross CS, Sadovnikoff N, Bader AM. Improving Preoperative Completion of Advanced Care Planning Documents in Patients With Expected Postoperative Intensive Care Unit Stay. A A Pract. 2019 Jun 15;12(11):455-458. doi: 10.1213/XAA.0000000000000993. PMID 30883399
- [Background] Hadler RA, Fatuzzo M, Sahota G, Neuman MD. Perioperative Management of Do-Not-Resuscitate Orders at a Large Academic Health System. JAMA Surg. 2021 Dec 1;156(12):1175-1177. doi: 10.1001/jamasurg.2021.4135. PMID 34550339
- [Background] Scally CP, Robinson K, Blumenthaler AN, Bruera E, Badgwell BD. Identifying Core Principles of Palliative Care Consultation in Surgical Patients and Potential Knowledge Gaps for Surgeons. J Am Coll Surg. 2020 Jul;231(1):179-185. doi: 10.1016/j.jamcollsurg.2020.03.036. Epub 2020 Apr 18. PMID 32311465